CLINICAL TRIAL: NCT00259350
Title: Prevention of Central Venous Catheter Infections : Comparison of the Efficacy of Skin Disinfection With 5% Povidone Iodine in Alcoholic Solution Versus 0.25% Chlorhexidine, 0.025 Benzalkonium and 4% Benzylic Alcohol
Brief Title: Chlorhexidine vs Povidone Iodine in Alcoholic Solutions for Prevention of Central Venous Catheter Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anticath
Record Dates: First submitted 2005-11-27; First posted 2005-11-29 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: ICU Patients Requiring a Central Venous Access
Keywords: Central venous catheter; Skin disinfection; Antisepsis; Nosocomial infection; Catheter infection
MeSH Terms: conditions — Cross Infection

INTERVENTIONS:
Drug: Skin disinfection

SUMMARY:
The best antiseptic solution for cateheter care remains unknown.High concentration in aquous solution or low concentration in alcoholic solution of chlorhexidine actbetter than povidone iodine in aquous solutions. No study has compare alcoholic formulations of low concentration of chlorhexidine and povidone iodine for skin disinfection prior to insertion of central venous catheters.

To compare the incidence of central venous catheter colonization after skin disinfection with either an alcoholic solution of povidone iodine or a combination of 0.5% chlorhexidine, 0.025% Benzalkonium and 4% benzylic alcohol.

To compare the incidence of catheter related bacteremia in the to study groups. To compare the local and general tolerance of the two antiseptic formulations

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 yeras of age
* Requiring an internal jugular or sub-clavian central venous catheter for their care during at least 72 h
* Informed consent signed up

Exclusion Criteria:

* Bacteriemic infection not under control
* extensive cutaneous infection
* Women with childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520
Dates: Start 2004-05; Study Completion 2006-04

PRIMARY OUTCOMES:
Prevention of catheter colonization

SECONDARY OUTCOMES:
Prevention of catheter related bacteremia
Prevention of a positive culture of the catheter whaterver the threshold
Local and general tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MIMOZ, MD, PhD, Study Chair — University Hospital of Poitiers, france
Locations (1):
- University hospital, Poitiers, Vienne, France

REFERENCES:
- [Derived] Mimoz O, Villeminey S, Ragot S, Dahyot-Fizelier C, Laksiri L, Petitpas F, Debaene B. Chlorhexidine-based antiseptic solution vs alcohol-based povidone-iodine for central venous catheter care. Arch Intern Med. 2007 Oct 22;167(19):2066-72. doi: 10.1001/archinte.167.19.2066. PMID 17954800